CLINICAL TRIAL: NCT04402814
Title: Evaluation and Correlation of SARS-Cov2 Virus IgG/IgM Rapid Test Cassette Clungene Test With the Standard Method of COVID19 Testing in Inpatients With or Without COVID19
Brief Title: IgG/IgM Antibody Test in Patients Who Have Tested Negative or Positive for COVID-19 With the Standard Method of COVID19 Testing.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fadi Haddad, M.D. (Other)
Responsible Party: Sponsor-Investigator, Fadi Haddad, M.D., Infectious Disease Specialist, Sharp HealthCare
Organization: Sharp HealthCare (Other)
Other Study IDs: IgG/IgM COVID19; 2005801 (Other: Sharp HealthCare Institutional Review Board (SHC IRB))
Record Dates: First submitted 2020-05-22; First posted 2020-05-27 (Actual); Last update posted 2020-07-27 (Actual); Status verified 2020-07

CONDITIONS: SARS-CoV 2
Keywords: Coronavirus; COVID-19; Clungene; IgG/IgM antibodies
MeSH Terms: conditions — Coronavirus Infections; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Arm A (positive for COVID-19): One or two samples of your blood that were previously collected for routine care will be obtained from the hospital laboratory and will be tested for the antibodies against COVID-19 virus.
  * First blood sample obtained: 7 to 12 days following onset of symptoms; and/or
  * Second blood sample obtained: 12 to 40 days following the onset of symptoms.
  Interventions: Diagnostic Test: Clungene rapid test cassette
- Arm B (negative for COVID-19): One sample of blood that was collected for routine care at any point during hospitalization will be obtained from the hospital laboratory and will be tested for the antibodies.
  Interventions: Diagnostic Test: Clungene rapid test cassette

INTERVENTIONS:
Diagnostic Test: Clungene rapid test cassette — Blood will be tested for the presence of IgG and IgM antibodies using the Clungene rapid test cassette.

SUMMARY:
The purpose of this study is to evaluate point of care SARS-Cov2 Virus IgG/IgM rapid test cassette Clungene test and correlate it with the standard method of testing in inpatients who have tested positive or negative for COVID19.

DETAILED DESCRIPTION:
This is a laboratory testing study using the SARS-Cov2 Virus IgG/IgM rapid test cassette Clungene test to determine the presence of IgM and IgG antibodies in subjects who have tested negative or positive for COVID-19. The study is observational and subjects will be assigned to one of two arms depending on the results of their nCOVID-19 test.

ELIGIBILITY:
Inclusion Criteria:

* Received confirmed COVID-19 positive or negative test from Sharp HealthCare's standard method of testing.
* Age >/=18 years old.
* Access to a phone in the hospital room or an electronic device that is capable of receiving phone calls and/or video calls and/or e-mail.
* Able to read/write/speak English or Spanish fluently.
* Subjects must have the ability to understand the requirements of the study, provide informed consent, and provide authorization of use and disclosure of personal health information.
* Hospitalized at the time of consent or recently discharged with leftover blood stored at hospital laboratory

Exclusion Criteria:

* Impaired cognitive or decision-making capacity (based on the clinical judgment of the PI or designee)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized (or recently discharged) subjects who have been previously tested for COVID-19 with the standard method of testing.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2020-05-05 (Actual); Primary Completion 2020-10-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
IgG/IgM antibodies | from date of consent to date of test completion, up to 40 days
  Presence of IgG and/or IgM antibodies

CONTACTS AND LOCATIONS:
Overall Officials: Fadi Haddad, MD, Principal Investigator — Sharp HealthCare
Locations (3):
- United States (3):
  - Fadi A. Haddad MD Inc., La Mesa, California
  - Sharp Grossmont Hospital, La Mesa, California
  - Sharp Memorial Hosptial, San Diego, California

IPD SHARING:
Plan to Share IPD: No